CLINICAL TRIAL: NCT06318026
Title: Systematic Implementation of Patient-centered Care for Alcohol Use Trial: Beyond Referral to Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01AA031231 (NIH); R01AA031231 (NIH)
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Unhealthy Alcohol Use
Keywords: Patient-centered care; Shared decision-making; Population-based management; Quality improvement; Decision aid
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: EHR and survey (latter masked)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Centralized Intervention (Experimental): A centralized intervention by a social worker or counselor, added to usual care that systematically offers outreach and shared decision-making for symptoms due to alcohol use.
  Interventions: Behavioral: Centralized Intervention
- Primary Care Intervention (Experimental): A primary care intervention added to usual care that uses state-of-the-art implementation interventions to systematically encourage primary care providers to offer routine shared decision-making for symptoms due to alcohol use.
  Interventions: Other: Primary Care Intervention
- Usual Care (No Intervention): Usual primary care

INTERVENTIONS:
Behavioral: Centralized Intervention — A centralized intervention by a social worker or counselor, added to usual care that systematically offers outreach and shared decision-making for symptoms due to alcohol use
  Arms: Centralized Intervention
Other: Primary Care Intervention — A primary care intervention added to usual care that uses state-of-the-art implementation interventions to systematically encourage primary care providers to offer routine shared decision-making for symptoms due to alcohol use.
  Arms: Primary Care Intervention

SUMMARY:
The Systematic Implementation of Patient-centered Care for Alcohol Use Trial is a pragmatic, cluster-randomized, effectiveness-implementation trial testing two interventions in Kaiser Permanente Washington to systematically implement shared decision-making with primary care patients with symptoms due to alcohol use: a primary care intervention and a centralized intervention. An anticipated 25 primary care clinics will be randomized to one of three conditions: usual care or the primary care or centralized interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult primary care patients ≥18 years old on the day of a primary care appointment; and
2. ≥4 symptoms on the Alcohol Symptom Checklist, or 2-3 symptoms on the Alcohol Symptom Checklist with at least one symptom associated with high risk of progression to severe symptoms, documented in the electronic health record associated with the primary care appointment; and
3. high-risk drinking on the alcohol screening questionnaire (AUDIT-C ≥7) on the day of the Alcohol Symptom Checklist or in the prior 30 days documented in the electronic health record.

Exclusion Criteria:

1. Documented request to not participate in research, or
2. Patient was eligible for the Vanguard pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Documentation of alcohol or substance use disorder treatment in the electronic health record (including insurance claims). | Treatment initiated up to 12 months.
Continuous measure of change in alcohol use as documented on the AUDIT-C screening questionnaire. | Up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Bradley, MD, MPH, Principal Investigator — Kaiser Permanente; Gwen Lapham, PhD, MPH, MSW, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States